CLINICAL TRIAL: NCT02042313
Title: Postoperative Pain Management After Minimally Invasive Esophagectomy
Acronym: MIEPVBEA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Nai Liang Li, MD, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20131015A
Record Dates: First submitted 2014-01-15; First posted 2014-01-22 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Epidural (Active Comparator): Epidural catheters will be applied at the T6-8 level prior to the induction. 6 ml of 2% xylocaine with 1 in 200,000 epinephrine administered before surgery. During the surgery, 2% xylocaine with 1 in 200,000 epinephrine infusion will be administered at a rate of 2-10 ml/hour adjusted according to patient's blood pressure. After surgery, 0.125% levobupivacaine with 2.5μg fentanyl and 1 in 400,000 epinephrine will be given at a rate of 0.10-0.15 ml kg-1 h-1 (0.5 h lock and 2 ml bolus) through a patient-controlled infusion pump.
  Interventions: Other: continuous epidural infusion
- combined PVB TAP (Experimental): Paravertebral catheterization into the paravertebral region ipsilateral to the VATS incision as described by Murata at the level of T7-8 will be performed. 10 ml of 2% xylocaine with 1 in 200,000 epinephrine to initiate analgesia. During the surgery, 2% xylocaine with 1 in 200,000 epinephrine infusion will be administered at a rate of 2-10 ml/hour adjusted according to patient's blood pressure. After the surgery, 0.125% levobupivacaine with 2.5μg fentanyl and 1 in 400,000 epinephrine will be administered at the rate of 0.10-0.15 ml kg-1 h-1 (0.5 h lock and 2 ml bolus) through a patient-controlled infusion pump.
  Ultrasound-guided (USG) subcostal TAP block will be performed at the end of surgery. Fifteen milliliters of 0.5% levobupivacaine with 1 in 400,000 epinephrine will be injected in incremental doses on each side of the abdomen.
  Interventions: Other: combined paravertebral infusion and single shot of TAP block

INTERVENTIONS:
Other: continuous epidural infusion
  Arms: Epidural
Other: combined paravertebral infusion and single shot of TAP block
  Arms: combined PVB TAP

SUMMARY:
Esophagectomy is a major surgical procedure often associated with significant morbidity and mortality and significant level of postoperative pain. In contrast to open esophagectomy where epidural pain control has been considered as a gold standard and could be crucial in affecting outcome the analgesic scheme for minimally invasive esophagectomy (MIE) is yet to be established. We would like to compare continuous epidural analgesia and continuous paravertebral block combined with single shot subcostal transversus abdominis plane (TAP) block in the analgesic effects, levels of cytokines, and postoperative complications in patients receiving MIE.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a physical status between ASA I and III
* 20 - 75 years of age
* Patient has signed an informed consent
* Without contraindication of GA, EA or PVB

Exclusion Criteria:

* ASA > III
* Inability to provide informed consent
* Bleeding disorders
* Being pregnant
* Contraindications to nonsteroidal anti-inflammatory drugs (NSAIDs),
* Allergy to amide-type local anesthetics or NSAIDs
* Infection at the thoracic paravertebral injection site
* Severe spine or chest wall deformity
* Patients with major psychosis or drug and alcohol abuse
* Patients with a history of significant neurological, psychiatric, neuromuscular, cardiovascular, pulmonary, renal or hepatic disease
* Patients with physical disability that precludes complete cooperation

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Intraoperative hypotension ( > 30% decline in the preoperative systolic/diastolic blood pressure) | during operation

SECONDARY OUTCOMES:
NRS pain score | postoperative day 0 to 4

OTHER OUTCOMES:
Tidal volume | postoperative day 1 to4

CONTACTS AND LOCATIONS:
Locations (1):
- Koo Foundation Sun Yat-Sen Cancer Center, Taipei, Taiwan, Taiwan